CLINICAL TRIAL: NCT04872387
Title: Randomized, Placebo-controlled, Single-blind, Dose Escalation Study to Investigate the Safety, Tolerability, and Pharmacokinetics After Single and Multiple Nasal Doses of BAY 2586116 in Japanese Healthy Male Participants
Brief Title: A Study to Learn More About How Safe BAY2586116 is, How it Affects the Body, How it Moves Into, Through and Out of the Body at Different Doses in Healthy Japanese Male Participants After Taking Single and Multiple Doses Through the Nose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: 20906
Record Dates: First submitted 2021-04-30; First posted 2021-05-04 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Phase I study; Japanese healthy volunteer study
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAY2586116 Dose step 1 and Placebo (Experimental): Each participant of Dose step 1 will receive a single dose of BAY2586116 or placebo.
  In this dose step, 12 participants will be included (9 on active treatment, 3 on placebo).
  Interventions: Drug: BAY2586116; Drug: Placebo
- BAY2586116 Dose step 2 and Placebo (Experimental): Each participant of Dose step 2 will receive a single dose of BAY2586116 or placebo.
  In this dose step, 12 participants will be included (9 on active treatment, 3 on placebo).
  Interventions: Drug: BAY2586116; Drug: Placebo
- BAY2586116 Dose step 3 and Placebo (Experimental): Each participant of Dose step 3 will receive single and multiple doses of BAY2586116 or placebo administered once daily (OD) for 5 consecutive days.
  In this dose step, 12 participants will be included (9 on active treatment, 3 on placebo).
  Interventions: Drug: BAY2586116; Drug: Placebo

INTERVENTIONS:
Drug: BAY2586116 — Nasal administration
Drug: Placebo — Matching placebo

SUMMARY:
BAY2586116 is a new drug in development for the treatment of obstructive sleep apnea. This is a condition that causes breathing to repeatedly stop and start during sleep due to blocked upper airways.

This is a study to learn more how safe BAY2586116 is, how it affects the body, how it moves into, through and out of the body in healthy Japanese male participants.

The participants will be randomly chosen to receive 1 of 3 different doses of BAY2586116 or to receive a placebo. A placebo looks like a treatment but does not have any medicine in it. The participants will receive their study treatment either 1 single time or once a day for 5 days through a nasal spray.

The participants will be in the study for a total of about 12 weeks. They will stay at their study site for either 5 or 9 days, depending on which study treatment they receive. During this time, the doctors will take blood and urine samples and check the participants' health. About 6 to 8 days after the participants receive their last treatment, the researchers will check the participants' health again.

The main aim of this study is to learn more about how safe BAY2586116 is compared to the placebo. To answer this question, the researchers will count the number of participants who have medical problems that may or may not be related to the study treatment. These medical problems are also known as "adverse events" while they are in the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation (including medical and surgical history, physical examination, laboratory tests, ECG, vital signs).
* Participant must be 20 to 45 years of age inclusive, at the time of signing the ICF.
* BMI above or equal 18.0 and below or equal 29.9 kg/m² at screening.
* Male.
* Japanese.
* Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* A sexually active man who has not been surgically sterilized has to agree not to act as sperm donor for the time period between signing of the ICF and 90 days after the last administration of study intervention.

Key Exclusion Criteria:

* A history of relevant diseases of vital organs, of the CNS (central nervous system) or other organs.
* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study intervention will not be normal.
* Given the nasal administration route, these diseases include (but are not limited to) any symptomatic and/or a history of relevant diseases of the ear, nose, and throat area (e.g. acute allergic rhinitis, acute infectious rhinitis, acute or chronical sinusitis, infection of the upper respiratory tract, symptomatic deviation of the nasal septum or a different relevant impairment of nasal breathing, history of any surgery of the ear, nose, and throat area [exception: sole history of adenectomy and/or tonsillectomy and/or paracentesis >1 year prior to 1st administration of study intervention], anatomical abnormalities of the ear, nose, and throat area [e.g. surgical corrected or uncorrected cheilognathopalatoschisis]).
* Liver insufficiency or active liver disease, which may include unexplained persistent transaminase elevations.
* Known or suspected liver disorders (e.g. Morbus Gilbert/Meulengracht) and bile secretion/flow (cholestasis, also history of it).
* Participants with thyroid disorders as evidenced by assessment of thyroid stimulating hormone levels outside the normal reference range at screening.
* Personal or familial history of genetically muscular diseases.
* History of autoimmune disease.
* Known hypersensitivity to the study interventions (active substances or excipients of the preparations).
* Known severe allergies, e.g. allergies to more than 3 allergens, allergies affecting the lower respiratory tract, allergic asthma, allergies requiring therapy with corticosteroids, urticarial, or significant non-allergic drug reactions.
* History of known or suspected malignant tumors.
* Tendency for vasovagal reactions (e.g. after venipuncture) or history of syncope.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From first administration up to 8 days after last dose (follow-up visit)

SECONDARY OUTCOMES:
Cmax of BAY2586116 | Day 1
  Cmax: maximum observed drug concentration in measured matrix after single dose administration.
Cmax/D of BAY2586116 | Day 1
  Cmax/d: Cmax divided by dose.
AUC of BAY2586116 | Day 1
  AUC: area under the concentration vs. time curve from zero to infinity after single (first) dose.
AUC/D of BAY2586116 | Day 1
  AUC/D: AUC divided by dose.
Cmax,md of BAY2586116 | Day 5
  Only for Dose step 3.
Cmax,md/D of BAY2586116 | Day 5
  Only for Dose step 3.
AUCτ,md of BAY2586116 | Day 5
  Only for Dose step 3. AUCτ,md: AUC during any planned dose interval after multiple dose.
AUCτ,md/D of BAY2586116 | Day 5
  Only for Dose step 3. AUCτ,md/D: AUCτ,md divided by dose.

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field — http://clinicaltrials.bayer.com/